CLINICAL TRIAL: NCT03752710
Title: Biometric Indicators of Eyes With Occult Lens Subluxation
Brief Title: Biometry of Occult Lens Subluxation Misdiagnosed as Primary Acute Angle Closed Glaucoma
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Principal Investigator, Lv Yingjuan, Dr Lv Yingjuan, Tianjin Medical University Eye Hospital
Other Study IDs: Tianjin LS study
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Subluxation of Lens
MeSH Terms: conditions — Lens Subluxation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Acute primary angle closure
- Acute secondary angle closure induced by LS
- Cataract
- Primary chronic angle closed glaucoma

SUMMARY:
In this work, we evaluated the biometry data of lens subluxation inducing acute angle closure which were misdiagnosed as primary angle closure at the first visit, and compared with the data of chronic angle closure glaucoma, cataract, primary acute angle closure.

ELIGIBILITY:
ASAC-LS was diagnosed according to the following criteria, including sudden pain in the eye, decreased vision with or without nausea and vomiting. Slit lamp microscopy reveals phacodonesis, lens inclination or vitreous herniation into the anterior chamber, central and peripheral shallow anterior chamber, and asymmetric iris bulge. All patients were confirmed during the surgery to have LS.

APACG was diagnosed with the following criteria6, 7 8, including substantially elevated IOP and closed angle, acute eye pain, blurred vision, or nausea and vomiting. More importantly, ischemic injury caused by acute ocular hypertension, ciliary or mixed congestion, corneal edema, and glaucoma flecks should be detected.

The diagnostic criteria of CPACG included narrow angle with anterior synechiae of varying widths, IOP > 22 mmHg, and glaucomatous optic disc damage and visual field shrinkage9-11 The angle closure should be more than two quadrants, yet there was no ischemic injury in the anterior segment caused by acute ocular hypertension.

Exclusion criteria were history of laser peripheral iridotomy or peripheral iridectomy, glaucoma filtration surgery, angle closure caused by ocular trauma, uveitis, neovascularization or lens swelling or hyper mature lens. The patients with acute angle closure in both eyes were excluded. The subjects in which Lenstar LS900 examination could not be performed because of severe lens opacity or corneal edema were also not included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective case study included 17 eyes of 17 patients with ASAC-LS, who were misdiagnosed with APACG on their first visit. In addition, 56 eyes of 56 patients diagnosed with APACG, 54 eyes of 54 patients diagnosed with CPACG, and 56 eyes of 56 patients diagnosed with cataract were also included. All of the patients were admitted from Jan 10, 2016 to Dec 28, 2017 in Tianjin Medical University Hospital. This study was conducted in accordance with the Helsinki Declaration and was approved by the Ethics Committee of Tianjin Medical University Eye Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Eye anterior segment biometry | 1 day
  Anterior segment biometry measure by Lenstar LS900
Intraocular pressure | 1 year
  Intraocular pressure was measured by Goldmann tonometer
visual acuity | 1 year
  visual acuity before and after surgery

REFERENCES:
- [Derived] Xing X, Huang L, Tian F, Zhang Y, Lv Y, Liu W, Liu A. Biometric indicators of eyes with occult lens subluxation inducing secondary acute angle closure. BMC Ophthalmol. 2020 Mar 5;20(1):87. doi: 10.1186/s12886-020-01355-7. PMID 32138781